CLINICAL TRIAL: NCT06130722
Title: First-in-Human, Phase I, Open-label, Multicenter, Dose Escalation Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of FL115 Monotherapy in Patients With Locally Advanced/Metastatic Solid Tumors
Brief Title: First-in-Human, Phase I, Open-label, Multicenter, Dose Escalation Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Forlong Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL115-101
Record Dates: First submitted 2023-11-07; First posted 2023-11-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: Open-label, Multicenter, Dose escalation Clinical Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A Single Arm (Experimental)
  Interventions: Drug: FL115

INTERVENTIONS:
Drug: FL115 — FL115 is a novel long-acting IL-15 agonist designed as a fusion protein with a mutated IL-15 structure (IL-15[N72D]/IL-15Rα-sFc).

SUMMARY:
First-in-Human, Phase I, open-label, multicenter, dose-escalation study to evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of FL115 in patients with advanced solid tumors who have progressed or are intolerant to current standard-of-care therapies, including immune check-point inhibitors administered in single-agent or combination use.

DETAILED DESCRIPTION:
This is a First-in-Human, Phase I, open-label, multicenter, dose-escalation clinical study to evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of FL115 when administered IV to adult patients with locally advanced/metastatic solid tumors who have progressed on, cannot tolerate, or do not have a standard-of-care therapy. If a patient is intolerant to standard-of-care therapy, the reason that the treatment could not be tolerated will be documented in the electronic case report form (eCRF). Patients will receive the investigational drug FL115 on Days 1, 8, 15, and 22 of Cycle 1 for the observation of AEs/SAEs to assess dose-limiting toxicity (DLT) in first 28 days. FL115 will be administered IV QW (on Days 1, 8, 15, and 22) in Cycle 2 and beyond. All patients will be monitored in the clinic over 24-hours for the C1D1 dose for monitoring potential cytokine release syndrome (CRS). If no CRS symptoms are observed after first dose, patients will not be asked for 24-hour inpatient monitoring for future injections (i.e. 2nd, 3rd and 4th dosing) based on the investigator discretion.

Seven dosing cohorts are planned, with doses of 3, 10, 30, 60, 120, 180 and 240 µg/kg.

For ethical reasons, the first 2 dose cohorts (3 and 10 µg/kg) are planned to enroll 1 patient per cohort because these 2 doses are considered suboptimal treatment for late-stage cancer patients. The first 2 dose level cohorts will each enroll 1 patient using an accelerated titration dose escalation design. If no DLT is observed by the end of the first cycle (28 days) of treatment, the dose will be escalated to the next dose cohort. However, if 1 treatment-related National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) or American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading ≥ Grade 2 toxicity occurs in the safety evaluation window, the study will be converted to a 3 + 3 design. After the initial 2 cohorts are completed, the study will use modified Fibonacci 3 + 3 dose-escalation design.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures
3. Histologically or cytologically confirmed incurable, unresectable, locally advanced or metastatic cancer that is refractory to standard therapies
4. Prior therapy:

   • Progressed on or are intolerant to all standard therapies including checkpoint inhibitors (such as PD-1, PDL-1, CTLA-4) as a single agent or in combination with oncolytic vaccine, antibody, or chemotherapeutic agents
5. Patient has at least 1 measurable target lesion or evaluable disease according to RECIST version 1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Patient's life expectancy ≥ 6 months
8. Adequate hepatic function as evidenced by meeting all of the following requirements:

   * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN); or ≤ 5 × institutional ULN for patients who have serum bilirubin increases due to underlying Gilbert's Syndrome (familial benign unconjugated hyperbilirubinemia).
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 2.5 × ULN; AST or ALT ≤ 5 × ULN if liver metastases are present
9. Adequate renal function as serum creatinine < 1.5 × ULN and calculated creatinine clearance (CrCL) ≥ 60 mL/min (Cockcroft-Gault Equation).
10. Hematological function defined as:

    * Absolute neutrophil count ≥ 1,500/µL without growth factor support in the 2 weeks prior to study entry
    * Hemoglobin > 9 g/dL without transfusion in the 2 weeks prior to study entry
    * Platelet count ≥ 100,000/µL without transfusion in the 2 weeks prior to study entry
11. Prothrombin (PT), international normalized ratio (INR), or activated partial thromboplastin time (aPTT) < 1.5 × ULN; use of full dose anticoagulants is permitted. These laboratory test values should be maintained within the therapeutic range and closely monitored by the Investigator.
12. Female patients of childbearing potential and male patients with partners of childbearing potential agree to use a highly effective form(s) of contraception during study treatment that results in a low failure rate of < 1% per year when used consistently and correctly. Male patients must always use a condom. Female patients of reproductive potential must not be pregnant, breastfeeding, or planning to conceive children within the duration of the study, beginning at the Screening visit (Initial Visit) through 120 days or for an additional 5 half-lives after the last dose of study treatment, whichever is longer. For female patients of reproductive potential, confirmation that the patient is not pregnant must be obtained by a negative serum pregnancy test result obtained during Screening.

    Note: Women will not be considered in the category of 'female patients of reproductive potential' if they have undergone surgical sterilization (including hysterectomy, bilateral oophorectomy or total hysterectomy), or who are postmenopausal (defined as no menses for more than 12 consecutive months without medical interference). Highly effective methods of contraception include combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only 1 partner during the whole study duration), and sexual abstinence. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug.
13. Able to stay in a 24-hour inpatient unit after 1st infusion visit and subsequent dosing visits as needed.

Exclusion Criteria:

1. Prior major surgery, chemotherapy, immunotherapy, or radiation therapy within 14 days prior to initiation of study treatment. No AE is evident from prior anticancer therapy except Grade 2 alopecia, sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement. Palliative radiotherapy to a single area of metastasis is allowed (consult with assigned Medical Monitor)
2. Prior allogeneic stem cell, bone marrow, or solid organ transplant.
3. Live virus vaccine within 30 days prior to study entry
4. Known active autoimmune disease or history of autoimmune disease requiring systemic therapy within 2 years prior to entry; except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type 1 diabetes mellitus
5. Use of systemic corticosteroids in a dose equivalent to > 10 mg/day of prednisone or other immunosuppressive agent within 2 weeks prior to study entry. Use of inhaled, topical, or ophthalmological steroids are allowed
6. Symptomatic CNS metastases. Patients with asymptomatic CNS metastases who are radiologically and neurologically stable ≥ 4 weeks following CNS directed therapy and are on a stable or decreasing dose of corticosteroids (e.g., prednisone less than 10 mg/day or equivalent) are eligible for study entry
7. Uncontrolled hypertension (systolic blood pressure > 160 mmHg and diastolic blood pressure > 99 mmHg), with symptoms or a known history of hypertension crisis, or hypertensive encephalopathy
8. Severe cardiovascular disease, including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction, or unstable angina within 6 months of study entry; New York Heart Association (NYHA) class III or IV heart failure within 6 months of study entry; uncontrolled arrhythmia within 6 months of study entry
9. Resting QTcF interval > 470 msec on ECG at baseline; no concomitant medications that would prolong the QT interval; known family history of long QT syndrome. Left ventricular ejection fraction <40% at baseline.
10. Concurrent malignancy within 2 years except cervical carcinoma in situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer under active surveillance, ductal carcinoma in situ of the breast, or ≤ T1 urothelial carcinoma
11. Known active infection including HIV, hepatitis B or C, or tuberculosis, requiring active therapy; exceptions are as follows:

    * Patients infected with the HIV virus will be eligible if their CD4 count is > 350 cells/mm3 and the patient is on anti-retroviral therapy with an HIV viral load that is below the level of detection.
    * Active Hepatitis B or C. HBV carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL), or inactive Hepatitis C (negative HCV RNA test) may be enrolled.
12. Known or suspected hypersensitivity to FL115 or its excipients; known history of a Grade 3 or 4 allergic reaction to IL treatment or another fusion protein.
13. Women of childbearing potential who do not consent to use 2 highly effective methods of birth control (including 1 barrier method) during treatment and for an additional 5 half-lives or 120 days after the last administration of study drug, whichever is longer.
14. Men with a partner of childbearing potential who do not consent to use 2 highly effective methods of birth control (including 1 barrier method) during treatment and for an additional 5 half-lives or 120 days after the last administration of study drug, whichever is longer.
15. Any condition that the Investigator or primary physician believes may not be appropriate for the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of FL115 in approximately 26 patients with unresectable locally advanced or metastatic solid tumors | From screening to 30 days after last dose.
  The study eligible patients will receive the investigational drug FL115 on Days 1, 8, 15, and 22 of Cycle 1 for the observation of AEs/SAEs to assess dose-limiting toxicity (DLT) in first 28 days. FL115 will be administered IV QW (on Days 1, 8, 15, and 22) in Cycle 2 and beyond. All patients will be monitored in the clinic over 24-hours for the C1D1 dose for monitoring potential cytokine release syndrome (CRS). If no CRS symptoms are observed after first dose, patients will not be asked for 24-hour inpatient monitoring for future injections (i.e. 2nd, 3rd and 4th dosing) based on the investigator discretion. Adverse events (AEs) and serious adverse events (SAEs), other than those associated with CRS and related neurotoxicity events, will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - HOAG Memorial Hospital Presbyterian, Newport Beach, California
  - Moores Cancer Center at UCSD Health, San Diego, California
  - Gabriel Cancer Center, Canton, Ohio